CLINICAL TRIAL: NCT04964596
Title: Managing Colorectal Cancer Prevention Procedure Wait Lists During the COVID-19 Pandemic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was never started due to lack of staff
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 21.210
Record Dates: First submitted 2021-07-09; First posted 2021-07-16 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Adenomatous Polyps
Keywords: Polyps detection; triage approach
MeSH Terms: conditions — Adenomatous Polyps | interventions — Colonoscopy; Colonography, Computed Tomographic

STUDY DESIGN:
Intervention Model Description: patients who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1:1 ratio into 3 groups
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- a colonoscopy as surveillance exam (Active Comparator): patients will undergo Colonoscopy, finding will be documented. Findings of colonoscopy will be documented and treated according to the institutional standards. Study participation for patients ends after the colonoscopy and follow-up of pathology results and complication assessment.
  Interventions: Diagnostic Test: colonoscopy
- undergoing a FIT as surveillance exam (Active Comparator): if the FIT test is positive: patients will have subsequent colonoscopy within 3 months. Findings of FIT testing and if positive the colonoscopy will be documented and participation in the study will end after that. Findings of the FIT test and colonoscopy will be treated according to the institutional standards. If FIT test is negative patient will leave the study and will have a follow up with a colonoscopy or FIT test in 1 to 2 years outside of this study.
  Interventions: Diagnostic Test: FIT test
- undergoing CT colonography as surveillance exam (Active Comparator): If CTC is positive: patients will have subsequent colonoscopy within 3 months. Findings will be documented and participation in the study will end there. Findings of the colonoscopy will be addressed according to our institution's guidelines. If CTC is negative for polypoid lesions patient will leave the study and will have a follow up 5 years after with either a CTC or colonoscopy.
  Interventions: Diagnostic Test: CT colonography

INTERVENTIONS:
Diagnostic Test: colonoscopy — colonoscopy
  Arms: a colonoscopy as surveillance exam
Diagnostic Test: FIT test — faecal immunochemical test
  Arms: undergoing a FIT as surveillance exam
Diagnostic Test: CT colonography — noninvasive medical imaging technique that uses computed tomography to visualize the interior of the colon and rectum especially to screen for polyps or cancerous growths
  Arms: undergoing CT colonography as surveillance exam

SUMMARY:
The main objective of this study is to offer and evaluate an interim triage approach for patients waiting for surveillance colonoscopies. This will reduce the waiting period and the psychological stressors for our patients and from a scientific point of view allow us to compare the yield of findings for each approach.

DETAILED DESCRIPTION:
This study will randomize patients (with low-risk findings in the initial colonoscopy) waiting for a surveillance colonoscopy into a follow-up with either FIT, CT colonography or colonoscopy. This approach will speed up the time for an exam for our patients and allow us to gather important data on the yield of significant findings when using FIT vs CT colonography vs colonoscopy for the surveillance exam.

All patients with positive FIT or CT colonography results will undergo subsequent colonoscopy. 300 patients will be randomized to 1:1:1 into 3 groups:

Group 1: patients will undergo Colonoscopy, findings will be documented and their participation in the study will end there. The findings of the colonoscopy will be addressed according to the institution's guidelines.

Group 2 will undergo fit testing if the fit test is positive: patients will have a subsequent colonoscopy within 3 months. Findings will be documented and participation in the study will end there. The findings of the colonoscopy will be addressed according to our institution's guidelines. If Fit test is negative patient will leave the study and will have a follow-up colonoscopy in one year.

Group 3 will have CT colonography. If CTC is positive: patients will have a subsequent colonoscopy within 3 months. Findings will be documented and participation in the study will end there. The findings of the colonoscopy will be addressed according to our institution's guidelines. If CTC is negative for polypoid lesions, the patient will leave the study and will have a follow-up 5 years after with a control colonoscopy.

All CT colonography and FIT tests analysis for patients will be performed as per the standard of care. Patients with suspicious lesions in CT colonography and positive FIT results will be redirected for colonoscopy and prioritized as P3 (Meaning endoscopy has to be done within 3 months).

Polypectomy specimens will be sent for pathological examination according to the standard of care and institutional routine practice. Pathology results will be followed up.

ELIGIBILITY:
Inclusion Criteria:

- people with referral sheets for surveillance colonoscopies : meaning 3 or 5 years after the initial colonoscopy.

Exclusion Criteria:

* known or suspected acute diverticulitis
* ulcerative colitis
* Crohn's disease
* toxic megacolon
* acute abdominal pain
* familial polyposis syndrome
* coagulopathy
* poor general health (defined as an American Society of Anaesthesiologists class >3)
* patients presenting for emergency colonoscopies
* patients incapable of lying flat on their back for the duration of the CT colonography due CHF or other predispositions
* patients with a personal history of CRC
* patient undergoing colonoscopy for surveillance after EMR or ESD procedures
* patients diagnosed with a CRC or a metastatic cancer
* patients with a history of contrast allergies
* Patients referred for polypectomy

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Number of detection of neoplastic colon polyp | 12 months
  Number of patients with a neoplastic colon polyp detected during colonoscopy
Comparaison of neoplastic colon polyp number detected between CTC and colonoscopy | 12 months
  The number of neoplastic colon polyp detected with the CTC compare to the number of neoplastic colon polyp detected with colonoscopy

SECONDARY OUTCOMES:
Number of patients on the list having a positive or negative FIT test or CTC and diagnosed with advanced neoplasia, non-advanced CR neoplasia, CR cancerous and precancerous lesions on colonoscopy | 12 months
  Number of patients on the list having a positive or negative FIT test or CTC and diagnosed with advanced neoplasia, non-advanced CR neoplasia, CR cancerous and precancerous lesions on colonoscopy
Number of patients on the list having a CTC and diagnosed with advanced neoplasia, non-advanced CR neoplasia, CR cancerous and precancerous lesions on colonoscopy | 12 months
  Number of patients on the list having a CTC and diagnosed with advanced neoplasia, non-advanced CR neoplasia, CR cancerous and precancerous lesions on colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier Universitaire de Montréal, Montreal, Quebec, Canada